CLINICAL TRIAL: NCT05581927
Title: Modified Whole-Body Hypothermia for Neonates With Hypoxic-Ischemic Encephalopathy
Brief Title: Whole-Body Hypothermia for Neonates With Hypoxic-Ischemic Encephalopathy(HIE)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients were included
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Children's Hospital of Suzhou (Unknown); Women and Children's Hospital of Chongqing (Unknown); Women and Children's Hospital of Guangxi (Unknown); People's hospital of Guangyuan (Unknown)
Responsible Party: Principal Investigator, Chen Long,MD, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Whole-Body Hypothermia
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-10

CONDITIONS: Hypoxic- Ischemic Encephalopathy; Whole-Body Hypothermia; Brain Injury
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Injuries

STUDY DESIGN:
Intervention Model Description: one group was allocated to standard Whole-Body Hypothermia, another group was allocated to modified Whole-Body Hypothermia
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified Whole-Body Hypothermia (Experimental): patients were allocated to modified Whole-Body Hypothermia with normal base excess and blood pressure.
  Interventions: Device: modified Whole-Body Hypothermia
- standard Whole-Body Hypothermia (Active Comparator): patients were allocated to standard Whole-Body Hypothermia.
  Interventions: Device: standard Whole-Body Hypothermia

INTERVENTIONS:
Device: modified Whole-Body Hypothermia — patients were allocated to modified Whole-Body Hypothermia with normal base excess and blood pressure
  Arms: modified Whole-Body Hypothermia
Device: standard Whole-Body Hypothermia — patients were allocated to standard Whole-Body Hypothermia
  Arms: standard Whole-Body Hypothermia

SUMMARY:
Among term infants, hypoxic-ischemic encephalopathy due to acute perinatal asphyxia remains an important cause of brain injury in childhood. Infants with moderate encephalopathy have a 10 percent risk of death, and those who survive have a 30 percent risk of disabilities. Sixty percent of infants with severe encephalopathy die, and many, if not all, survivors are disabled. Whole-body hypothermia reduces the risk of death or disability in infants with moderate or severe hypoxic-ischemic encephalopathy.

DETAILED DESCRIPTION:
Reductions in brain temperature by 2°C to 5°C provide neuroprotection in newborn and adult animal models of brain ischemia.Brain cooling has a favorable effect on multiple pathways contributing to brain injury, including excitatory amino acids, the cerebral energy state, cerebral blood flow and metabolism, nitric oxide production, and apoptosis. Brain cooling is effective in reducing the extent of brain injury even when it is initiated up to 5.5 hours after brain ischemia in near-term sheep fetuses.But, epidemiological data showed that, in non-developed countries and areas,Whole-body hypothermia is related to the increased mortality and brain injury. The cause is unclear.

ELIGIBILITY:
Inclusion Criteria:

* pH of 7.0 or less or a base deficit of 16 mmol per liter or more in a sample of umbilical cord blood or any blood during the first hour after birth. If, during this interval,a pH was between 7.01 and 7.15, a base deficit was between 10 and 15.9 mmol per liter. or a blood gas was not available, additional criteria were required.

These included an acute perinatal event (e.g., late or variable decelerations, cord prolapse, cord rupture,uterine rupture, maternal trauma, hemorrhage, or cardiorespiratory arrest) and either a 10-minute Apgar score of 5 or less or assisted ventilation initiated at birth and continued for at least 10 minutes.

* equal to or more than 36 weeks

Exclusion Criteria:

* congenital malformation
* parents' refusal

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
death | 30 days
  neonates are dead during hospital
brain injury | 30 days
  neonates are diagnosed with brain injury

SECONDARY OUTCOMES:
the incidence of suspend of Whole-Body Hypothermia | within 3 days
  Whole-Body Hypothermia is suspended
the incidence of discharge according to the doctor's suggestion | 2-3 weeks
  neonates were discharged according to the doctor's suggestion
the incidence of intraventricular hemorrhage | 2-3 week
  intraventricular hemorrhage was diagnosed
the incidence of periventricular leukomalacia | within 30 days
  Periventricular leukomalacia is diagnosed
neurodevelopmental assessment | one month
  neurodevelopment is assessed using NBNA
neurodevelopmental assessment | 18-36 months
  neurodevelopment is assessed using Bayley scale

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China